CLINICAL TRIAL: NCT03905434
Title: Evaluation of Circulating Exosomal MicroRNAs as Surrogate Stroke-Clock in Acute Anterior Circulation Large Vessel Occlusion
Brief Title: Identification of microRNAs Involved in Cerebral Collateral Regulation
Acronym: microRNA
Status: Suspended | Type: Observational
Why Stopped: PI moved from OSU to VCU. Study is suspended pending credentialing and IRB approval at VCU.
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor
Other Study IDs: HM20025643; 2018H0199 (Other: Ohio State University)
Record Dates: First submitted 2018-10-09; First posted 2019-04-05 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Cerebrovascular Disorders
Keywords: Large vessel occlusion; Acute ischemic stroke; microRNA
MeSH Terms: conditions — Cerebrovascular Disorders; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — microRNA sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: A total of 15 healthy controls will be enrolled and miRNA samples will be collected
  Interventions: Genetic: miRNA sampling
- Stroke: A total of 30 acute stroke patients with large vessel occlusions will be enrolled.
  Interventions: Genetic: miRNA sampling

INTERVENTIONS:
Genetic: miRNA sampling — Blood samples for miRNA testing will be collected from all subjects (control and patients diagnosed with acute ischemic stroke)

SUMMARY:
Patients >18 years of age presenting to Ohio State Wexner Medical Center Emergency department with stroke symptoms, within 6 hours of last know well and found to have acute anterior circulation large vessel occlusion (LVO) will be included in this study. The purpose of this study is to evaluate the differential expression of exosomal microRNAs in patients with stroke due to acute LVO as compared to healthy controls. In addition, the investigators will also evaluate the differential expression of exosomal microRNA in patients with good vs poor collateral grade.

DETAILED DESCRIPTION:
Patients aged >18 years presenting to the Emergency Department at the Ohio State University (OSU) Wexner Medical Center with acute ischemic stroke will be screened. The investigators will include patients with anterior circulation acute ischemic stroke secondary to sudden acute large vessel occlusion (LVO). Healthy subjects will be used as controls to assess miRNAs specific to stroke population. Since hemodynamically significant preexisting stenosis may result in alteration of miRNA expression, the investigators will exclude patients with >50% stenosis of internal carotid artery (ICA), >50% stenosis of bilateral vertebral arteries as well as patients with moderate to severe intracranial atherosclerotic disease as seen in CT Angiogram (CTA) of the head and neck. To minimize confounders, patients with known moderate to severe peripheral vascular disease or symptomatic coronary artery disease with history of stent or coronary artery bypass graft will also be excluded. Prisoners and Pregnant women will be excluded from this study as well.Differential expression of exosomal microRNAs in patients with acute LVO compared to healthy controls will be evaluated. In addition, a Neuroradiologist will grade the cerebral collateral circulation as (i) good or (ii) poor, after carefully reviewing CTA and CT perfusion (CTP) studies in each patient using validated collateral scoring method. Thirty patients with large vessel occlusion will be enrolled in this study in addition to 15 healthy controls (n=45). Blood samples will be drawn at 4 different time points from symptom onset for each patient: (i) 0-6 hours, (ii) 6-12 hours, (iii) 12-24 hours and (iv) 5-7 days. Differential MiRNA expression will also be evaluated between the patients with varying collateral grades

As the process of collateral maturation likely begins shortly after hemodynamic changes induced by LVO, the investigators plan to collect the first sample within 0-6 hours. Three blood samples will be collected during the first 24 hours to increase the chances of capturing the miRNA expression profile at the beginning of the collateral remodeling process. miRNA profiles of these patients will then be analyzed and compared to healthy volunteers. In addition, comparison will be done between patients with good and poor cerebral collateral grade.We will analyze the miRNA profiles of these patients using methods described below.

Exosome Isolation and Characterization: Quantification of exosome number and size will be carried out using a NanoSight NS300 (Nanosight, UK) at the OSU CCC Analytical Cytometry Core as previously described. Briefly, exosomes will be isolated from cell-free plasma using Total Exosome Isolation Kit (Invitrogen) according to the manufacturer's instructions. Exosomes will be suspended in PBS buffer and stored at 4° C for up to 7 days. The exosome suspension will then be diluted to achieve a working concentration between 2 x 108 - 8 x 108 for use in the NanoSight NS300, after which exosomes will be counted and sized11.

Total RNA Isolation: Total RNA will be isolated from exosomes suspended in PBS using the Circulating Nucleic Acid Extraction Kit (Qiagen) as previously described12. DNA contamination will be mitigated through use of Qiagen's RNase-free DNase set. RNA will be concentrated and purified using the RNeasy MinElute Cleanup Kit (Qiagen) as described.

NanoString Assay: The multiplexed nanoString nCounter miRNA system (nanoString Technologies) at The Ohio State University CCC Genomics Shared Resource will be used for miRNA expression profiling as described12. Total RNA (100ng) isolated from exosomes will be used as input material. Small RNA samples will be prepared by ligating a specific DNA tag onto the 3'-end of mature miRNAs according to manufacturer's instructions (nanoString Technologies). These tags will normalize the melting temperatures of the miRNAs and provide identification for each miRNA species in the sample. Excess tags will be washed away, and the resulting material hybridized with miRNA:tag-specific nCounter reporter probes. Hybridized probes will then be purified and immobilized on a streptavidin-coated cartridge using the nCounter Prep Station (nanoString Technologies). The nCounter Digital Analyzer will be used to count individual fluorescent barcodes and quantify miRNA molecules present in each sample.

miRNA Expression Profile Normalization and Analyses: Quality control, normalization, and data analyses will be performed using nSolver 2.0 Analysis Software (nanoString Technologies) as previously described. Hierarchical clustering of miRNAs identified through the nanoString query will be conducted using dChip (v 1.3) software. Differentially expressed miRNAs in patients with good or poor collateral scores (as described above) will be defined by a greater than or less than 2-fold change using one-way analysis of variance (ANOVA) assay with a significance level of p<0.05 and with correction for false discover rate.

RT-PCR Validation of Exosomal miRNAs: Select miRNAs isolated from exosomes will be reverse transcribed using the miRCURY LNA Universal cDNA synthesis kit (Exiqon) according to the manufacturer's protocol as described previously. miRNAs will be quantified by real-time PCR using ExiLENT SYBR Green (Exiqon) on a Mx3000P qPCR platform, with expression normalized to a housekeeping reference (i.e. SNORD44).

ELIGIBILITY:
Inclusion criteria:

1. Age 18 years or older.
2. Diagnosis of Acute Ischemic Stroke secondary to LVO
3. LVO from presumed embolic source (<50% ICA)
4. CT perfusion/RAPID images showing salvageable penumbra (evaluated by PI)

Exclusion:

1. >50% stenosis of internal carotid artery
2. >50% stenosis of bilateral vertebral arteries.
3. Patients with moderate to severe intracranial atherosclerotic disease as seen in CTA of head and neck.
4. Known moderate to severe PVD or symptomatic CAD
5. Past medical history of stent or coronary artery bypass surgery
6. Prisoners
7. Pregnant women
8. Previous stroke within 30 days
9. Intracranial vascular malformation or evidence of moya-moya disease
10. Serious advanced or terminal illness per judgment of the investigator with life expectancy <1yr
11. Known allergy to iodine that precludes CTA or CTP studies
12. Presumed septic embolus or suspected bacterial endocarditis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged >18 years presenting to the Emergency Department at Ohio State Wexner Medical Center with acute ischemic stroke within 6 hours of last known well will be screened. The investigators will include patients with acute anterior circulation LVO as identified by CT Angiogram. Healthy subjects will be used as controls to assess differentially expressed miRNAs specific to stroke population.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2018-08-14 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
identification of differentially expressed microRNAs in patients with sudden acute anterior circulation large vessel occlusion, compared to healthy controls. | 2 years
  The investigators will identify and report the microRNAs differentially expressed in patients with acute large vessel occlusion compared to healthy controls.

SECONDARY OUTCOMES:
Identification of differentially expressed microRNAs in patients with good vs poor cerebral collateral circulation | 2 years
  differential expression of microRNAs in participants with good and poor collateral circulation will be assessed and reported

CONTACTS AND LOCATIONS:
Overall Officials: Shraddha Mainali, MD, Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No